CLINICAL TRIAL: NCT07354594
Title: Adaptive External Beam and Radioligand Radiotherapy for MEtaSTatic Castration Resistant Prostate Cancer (ARREST): a Phase II Registry-based RCT
Brief Title: External Beam and Radioligand Radiotherapy for mCRPC
Acronym: ARREST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026-13179
Record Dates: First submitted 2025-11-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Metastatic Castration-Resistant
Keywords: radiotherapy; radioligand therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC radioligand therapy (Active Comparator)
  Interventions: Radiation: SOC radioligand therapy only
- External beam added to radioligand radiotherapy (Experimental)
  Interventions: Radiation: external beam radiotherapy delivered between cycles of radioligand radiotherapy

INTERVENTIONS:
Radiation: external beam radiotherapy delivered between cycles of radioligand radiotherapy — external beam radiotherapy delivered between cycles of radioligand radiotherapy
  Arms: External beam added to radioligand radiotherapy
Radiation: SOC radioligand therapy only — soc radioligand therapy only
  Arms: SOC radioligand therapy

SUMMARY:
Introduction 177Lu-PSMA radioligand therapy (RLT) is an emerging option for metastatic castration-resistant prostate cancer (mCRPC). However, up to half of patients fail to show meaningful clinical benefit with this therapy. A dual-modality strategy seeks to increase dose via complementary external beam radiotherapy (EBRT) in underdosed tumor regions. We hypothesize that by combining both modalities (EBRT and RLT) in an hybrid, adaptive approach, we can safely improve skeletal related events when compared to standard-of-care (SOC) 177Lu-PSMA alone.

Methodology Adaptive EBRT and RLT for mCRPC (ARREST) is a pragmatic registry-based phase 2, multi-center randomized controlled trial within the PERa prospective cohort (NCT03378856) planned to activate in 2025. Patients who are receiving SOC 177Lu-PSMA with targetable metastatic burden identified on imaging suitable for EBRT will be eligible. One hundred and thirty eligible patients will be randomized 1:1 to receive either SOC 177Lu-PSMA therapy alone (maximum 6 cycles) or to combined 177Lu-PSMA plus EBRT boost. Patients in the experimental arm will undergo FDG-PET at study entry and SPECT-CT after each cycle of radioligand therapy. Lesions selected for EBRT boost will be selected based on a set of criteria that include estimated suboptimal dose absorbed from 177LuPSMA, lesions demonstrating low PSMA but high FDG update, symptomatic lesions, and those at high risk for skeletal-related events. Selected lesions will receive single-fraction EBRT. Dose prescribed will range from 6-12 Gy with the ideal goal of a combined total biological effective dose of ≥75 Gy (α/β = 1.4) with priority to dose limits for organs at risk. A maximum treatment time of 60 minutes is permitted for each EBRT boost treatment. Patients in the experimental arm that achieve complete response measured by 177Lu-SPECT-CT and PSA will pause ARREST and resume at progression. The primary endpoint is skeletal related events at 1 year. Secondary objectives include overal survival, 177Lu-SPECT-CT and PSA response, toxicity, and quality of life. The sample size is designed to detect a 12 month imporvement in the rate of skeletal related events with a HR 1.6, two-sided alpha of 0.1 and 80% power.

Conclusion ARREST is hypothesized to safely optimize tumor dose, offering a personalized hybrid approach that may lead to improved patient outcomes. In addition, this study will permit further understanding of these two distinct radiation delivery methods and their effect on tissues, thereby refining the relative biological effectiveness model for more precise treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Receiving 177Lu-PSMA for mCRPC
* ECOG 0-1
* Presence of a discernible metastatic burden suitable for EBRT
* Receiving bone protective therapy

Exclusion Criteria:

* no exclusions

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Skeletal Related Events | 12 months

SECONDARY OUTCOMES:
Adverse Events | 12 months
  CTCAE Grade 2+ events
Overall suvival | 24 months
PSA Response | week 12
  Proportion of patients achieving a >'50% PSA decline
CR/PR on SPECT-CT | After 3 cycles
Quality of Life Questionnaires | 12 and 24 months
  EORTIC QLQ-C30, PRO-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Menard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided